CLINICAL TRIAL: NCT04477200
Title: Phase 0/I Dose Escalation Study of Mycophenolate Mofetil Combined With Radiation Therapy in Glioblastoma
Brief Title: Mycophenolate Mofetil Combined With Radiation Therapy in Glioblastoma
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of Michigan Rogel Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: UMCC 2019.192; HUM00175785 (Other: University of Michigan); R37CA258346 (NIH)
Record Dates: First submitted 2020-07-14; First posted 2020-07-20 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-06

CONDITIONS: Recurrent Glioblastoma; Recurrent Gliosarcoma; Recurrent Astrocytoma, Grade IV; Newly Diagnosed Glioblastoma; Newly Diagnosed Gliosarcoma; Newly Diagnosed Astrocytoma, Grade IV
Keywords: recurrent Glioblastoma; recurrent Gliosarcoma; newly diagnosed Glioblastoma; newly diagnosed Gliosarcooma; Recurrent Astrocytoma, Grade IV; Newly Diagnosed Astrocytoma, Grade IV
MeSH Terms: conditions — Glioblastoma; Gliosarcoma | interventions — Mycophenolic Acid; Radiotherapy; Temozolomide

STUDY DESIGN:
Intervention Model Description: Phase 0 will include 8 participants; eligible participants from phase 0 may continue on to phase 1.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Phase 0 - Recurrent glioblastoma (GBM) / gliosarcoma (GS) (Experimental): Mycophenolate mofetil
  Interventions: Drug: Mycophenolate Mofetil; Procedure: Re-resection (as part of standard of care)
- Phase 1 - Recurrent GBM / GS (Experimental): Mycophenolate mofetil; radiation therapy
  Interventions: Radiation: Radiation Therapy; Drug: Mycophenolate Mofetil
- Phase 1 - Newly Diagnosed GBM / GS (Experimental): Mycophenolate mofetil; radiation therapy; temozolomide
  Interventions: Drug: Temozolomide; Drug: Mycophenolate Mofetil; Radiation: Radiation Therapy

INTERVENTIONS:
Drug: Mycophenolate Mofetil — 500-2000mg orally twice daily, one week prior to re-resection (2 participants at each of 4 dose levels: 500mg, 1000mg, 1500mg and 2000mg)
  Other Names: MMF
  Arms: Phase 0 - Recurrent glioblastoma (GBM) / gliosarcoma (GS)
Radiation: Radiation Therapy — 40.5 Gy in 15 fractions
  Other Names: RT
  Arms: Phase 1 - Recurrent GBM / GS
Procedure: Re-resection (as part of standard of care) — Re-resection or biopsy of tumor as part of standard of care
  Arms: Phase 0 - Recurrent glioblastoma (GBM) / gliosarcoma (GS)
Drug: Temozolomide — Temozolomide capsules are an approved oral chemotherapeutic drug for the treatment of adult patients with newly diagnosed GBM/GS concomitantly with radiotherapy and then as adjuvant treatment. The dosing and timing of temozolomide therapy will be determined as per standard-of-care for the individual patient by the treating oncologist.
  Other Names: TMZ
  Arms: Phase 1 - Newly Diagnosed GBM / GS
Drug: Mycophenolate Mofetil — 250-2000mg orally twice daily, one week prior to and concurrent with RT.
  Other Names: MMF
  Arms: Phase 1 - Recurrent GBM / GS
Drug: Mycophenolate Mofetil — 250-2000mg orally twice daily, one week prior to and concurrent with RT and cyclic chemotherapy with temozolomide.
  Other Names: MMF
  Arms: Phase 1 - Newly Diagnosed GBM / GS
Radiation: Radiation Therapy — 60 Gy in 30 fractions
  Other Names: RT
  Arms: Phase 1 - Newly Diagnosed GBM / GS

SUMMARY:
This is a phase 0/1 dose-escalation trial to determine the maximum tolerated dose of Mycophenolate Mofetil (MMF) when administered with radiation, in patients with glioblastoma or gliosarcoma.

DETAILED DESCRIPTION:
The goal of the Phase 0 component is to determine if MMF achieves active concentrations in brain tumors. Eight participants in Phase 0 will receive MMF for one week before undergoing an already planned biopsy or re-resection (surgical removal) of glioblastoma or gliosarcoma (GBM/GS). A small portion of the tumor, removed as part of clinical care, will be used for testing in this study. Sixty additional participants will be enrolled in the Phase 1 component of the trial (30 with recurrent GBM/GS and 30 with newly diagnosed GBM/GS). The goal of the Phase 1 component is to find the dose of MMF that works best without causing severe side effects (the maximum tolerated dose) when combined with radiation in recurrent GBM/GS and with radiation and chemotherapy in newly diagnosed GBM/GS. Participants in Phase 0 who meet the eligibility criteria for the Phase 1 component may participate in both phases.

ELIGIBILITY:
Inclusion Criteria:

* Glioblastoma or gliosarcoma (recurrent or newly diagnosed).
* Karnofsky Performance Status 60 or greater.
* Phase 0: Candidate for clinically indicated re-resection or biopsy of glioblastoma or gliosarcoma per treating physician(s).
* Phase 1, Recurrent: Candidate for clinically indicated re-irradiation of glioblastoma or gliosarcoma per treating physician(s) (No more than one prior course of radiation for GBM).
* Phase 1, Newly Diagnosed: Candidate for upfront standard of care chemoradiation for glioblastoma or gliosarcoma per treating physician(s), to start no earlier than 14 days post- operatively from last definitive surgery for glioblastoma or gliosarcoma (if more than one surgery done. Ex. biopsy prior to resection).
* ANC >=1,500 cells/mm^3 within 14 days prior to enrollment.
* Patient (men and childbearing age women) agrees to the use of highly effective contraception during study participation and for at least 6 weeks for female patients and 90 days for male patients after final MMF administration.
* Ability to understand and the willingness to sign a written informed consent.

Exclusion Criteria:

* Lack of histopathological diagnosis of the tumor.
* Gliomatosis cerebri pattern (tumor involving 3 or more lobes) of disease.
* Leptomeningeal disease.
* Use of bevacizumab within 8 weeks of study enrollment.
* Known history of HIV.
* Active hepatitis B or C infection.
* Active systemic or central nervous system (CNS) infection.
* Grade 4 lymphopenia (if ALC <0.5, patient must be on Pneumocystis jirovecii prophylaxis).
* Estimated CrCl < 25 ml/min.
* History of organ transplantation.
* Patients with known hypoxanthine-guanine phosphoribosyl-transferase deficiency.
* Serious intercurrent disease.
* History of allergic reaction or hypersensitivity to mycophenolate mofetil or mycophenolic acid or any component of the drug product; or medical contraindication for MMF per treating physician(s).
* Known immunosuppressive condition from autoimmune disease, immune deficiency syndrome, or chronic immunosuppressive therapy.
* Inability to undergo MRI brain with and without contrast.
* Pregnant or lactating women.
* Patients with known phenylketonuria.
* Phase 0: Patients undergoing biopsy who are deemed unlikely to have sufficient tissue to spare for research purposes (e.g., those whose tumors are in an eloquent brain location where all tissue taken must be used for diagnostic purposes).
* Phase I: Increase in steroid requirement within 7 days of study enrollment (stable or decreasing dose allowed).
* Phase I, Recurrent: Radiation within 6 months prior to study enrollment.
* Phase I, Recurrent: Surgery within 4 weeks of re-irradiation.
* Phase I, Newly Diagnosed: History of hypersensitivity reactions to temozolomide or any other ingredients in temozolomide and dacarbazine.
* Phase I, Newly Diagnosed: Prior chemotherapy or radiation therapy for glioblastoma or gliosarcoma.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2020-08-05 (Actual); Primary Completion 2025-01-06 (Actual); Study Completion 2027-11-05 (Estimated)

PRIMARY OUTCOMES:
Concentration of mycophenolic acid (MPA) in tumor tissue in Phase 0 participants | At 1 week
  The concentration of MPA (the active metabolite of mycophenolate mofetil [MMF]) in tumor tissue, measured by mass spectrometry on a continuous scale after one week of MMF administration.
  This measure includes all phase 0 participants.
Number of recurrent phase 1 participants who experience dose-limiting toxicities (DLTs) at each dose level | Up to 28 days following completion of MMF + RT (up to ~9 weeks)
  DLT will be defined based on the rate of drug related grade 3-5 adverse events experienced from the start of treatment with MMF and for up to 4 weeks after completion of MMF + radiation therapy (RT). Assessed using National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) version 5.0.
  This measure includes only phase 1 participants with recurrent GBM/GS.
Number of newly diagnosed phase 1 participants who experience dose-limiting toxicities (DLTs) at each dose level -- DLT1 period | Up to 28 days following completion of MMF + RT + TMZ (up to ~11 weeks)
  DLT will be defined based on the rate of drug related grade 3-5 adverse events experienced from the start of treatment with MMF and for up to 4 weeks after completion of MMF + RT + TMZ. Assessed using National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) version 5.0.
  This measure includes only newly diagnosed phase 1 participants.
Number of newly diagnosed phase 1 participants who experience dose-limiting toxicities (DLTs) at each dose level -- DLT2 period | During the first 2 cycles (8 weeks) of MMF with adjuvant TMZ (up to ~19 weeks)
  DLT will be defined based on the rate of drug related grade 3-5 adverse events experienced during the first 2 cycles (8 weeks) of MMF with adjuvant TMZ. (The first cycle of MMF with adjuvant TMZ begins 28 days post-RT.) These will be assessed using National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) version 5.0.
  This measure includes only newly diagnosed phase 1 participants.

SECONDARY OUTCOMES:
Concentrations of guanosine triphosphate (GTP) in tumor tissue in Phase 0 participants | After one week of MMF administration
  The concentrations of GTP in tumor tissue, measured by mass spectrometry on a continuous scale.
  This measure includes all phase 0 participants.
Adverse events associated with treatment in all Phase 1 Participants | Up to 28 days following completion of MMF + RT (up to ~9 weeks)
  Toxicities at each dose level will be tabulated, categorized by grade and attribution.
  This measure includes all phase 1 participants.
Adverse events associated with treatment in newly diagnosed phase 1 participants | Up to 28 days following completion of MMF with adjuvant temozolomide (up to ~15 months)
  Toxicities at each dose level will be tabulated, categorized by grade and attribution.
  This measure includes only newly diagnosed phase 1 participants.
Overall Response Rate in phase 1 participants with recurrent GBM/GS | Until study stops or death; up to approximately 3 years.
  Determined by modified Response Assessment for Neuro-Oncology (mRANO) criteria. The number and proportion of patients with progressive disease, stable disease, partial and complete response will be calculated for each dose level and overall.
  This measure includes only phase 1 participants with recurrent GBM/GS.
Median Progression Free Survival (PFS) in phase 1 participants with recurrent GBM/GS | Until study stops or death; up to approximately 3 years.
  PFS defined as time from date of registration to the date of documented progressive disease, other disease related therapy or death. Determined by mRANO criteria.
  This measure includes only phase 1 participants with recurrent GBM/GS.
Median Freedom from Local Progression (FFLP) in phase 1 participants with recurrent GBM/GS | Until study stops or death; up to approximately 3 years.
  FFLP defined as time from date of registration to the date of documented local progressive disease. Determined by mRANO criteria.
  This measure includes only phase 1 participants with recurrent GBM/GS.
Median Overall Survival (OS) in phase 1 participants with recurrent GBM/GS | Until study stops or death; up to approximately 3 years.
  OS defined as time from date of registration to date of death or last follow up. Determined by Kaplan Meier method.
  This measure includes only phase 1 participants with recurrent GBM/GS.

CONTACTS AND LOCATIONS:
Overall Officials: Nathan Clarke, MD, Principal Investigator — University of Michigan Rogel Cancer Center
Locations (1):
- University of Michigan Rogel Cancer Center, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zhao G, Newbury P, Ishi Y, Chekalin E, Zeng B, Glicksberg BS, Wen A, Paithankar S, Sasaki T, Suri A, Nazarian J, Pacold ME, Brat DJ, Nicolaides T, Chen B, Hashizume R. Reversal of cancer gene expression identifies repurposed drugs for diffuse intrinsic pontine glioma. Acta Neuropathol Commun. 2022 Oct 23;10(1):150. doi: 10.1186/s40478-022-01463-z. PMID 36274161